CLINICAL TRIAL: NCT05906212
Title: Use of Anterior Lens Capsule as a Spacer in the Deep Sclerectomy _ Phacoemulsification: A Randomized Clinical Trial
Brief Title: Anterior Lens Capsule as a Spacer in the Deep Sclerectomy _ Phacoemulsification
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammadali Javadi, MD, Head of Ophthalmic Research Center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14021
Record Dates: First submitted 2023-05-16; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Glaucoma; Cataract
MeSH Terms: conditions — Glaucoma; Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nonpenetrating deep sclerectomy&phacoemulsification&autotransplantation of anterior lens capsule (Experimental): The intervention group will be undergoing non-penetrating deep sclerectomy and phacoemulsification with the use of an autotransplantation of the human anterior lens capsule as the spacer in the intrascleral lake.
  Interventions: Procedure: Non-penetrating deep sclerectomy and phacoemulsification and autotransplantation of anterior lens capsule
- Non-penetrating deep sclerectomy and phacoemulsification (Active Comparator): The control group will be undergoing non-penetrating deep sclerectomy and phacoemulsification without any spacer.
  Interventions: Procedure: Non-penetrating deep sclerectomy and phacoemulsification

INTERVENTIONS:
Procedure: Non-penetrating deep sclerectomy and phacoemulsification and autotransplantation of anterior lens capsule — This group will be undergoing nonpenetrating deep sclerectomy and phacoemulsification with autotransplantation of anterior lens capsule.
  Arms: Nonpenetrating deep sclerectomy&phacoemulsification&autotransplantation of anterior lens capsule
Procedure: Non-penetrating deep sclerectomy and phacoemulsification — This group will be undergoing nonpenetrating deep sclerectomy and phacoemulsification alone.
  Arms: Non-penetrating deep sclerectomy and phacoemulsification

SUMMARY:
In this randomized clinical trial, patients with concomitant glaucoma and cataract candidate for non-penetrating deep sclerectomy (NPDS) and phacoemulsification (PE) and subtenon mitomycin injection will be enrolled. Patients will randomly be allocated to two groups ["NPDS and PE and autotransplantation of human anterior lens capsule (ALC)" and "NPDS and PE" alone]. Exclusion criteria will be the patients with prior ocular surgery, neovascular glaucoma, uveitis, or compromised ocular surface. The intervention group will be undergoing NPDS and PE with the use of an ALC as the spacer in the intrascleral lake. The control group will be undergoing NPDS and PE without any spacer. The primary outcome will be intraocular pressure measured on days 1, 3, 7, months 1, 3, 6, and 12. The secondary outcomes will be surgical success rate (complete and qualified), the number of glaucoma medications, best-corrected visual acuity, surgical complications, and the need for needling and laser goniopuncture measured at the same intervals. The complete success rate will be defined as intraocular pressure less than 18 mmHg with a 20 percent reduction without anti-glaucoma medication. The qualified success rate will be defined as intraocular pressure less than 18 mmHg with a 20 percent reduction with anti-glaucoma medication.

ELIGIBILITY:
Inclusion criteria

* Patients with concomitant uncontrolled glaucoma and significant cataract
* Progression in glaucoma despite medical treatment
* Age more than 18 years old

Exclusion criteria

* Prior ocular surgery
* Neovascular glaucoma or uveitic glaucoma
* Compromised ocular surface or insufficient conjunctiva

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-05-16 (Estimated); Study Completion 2024-06-16 (Estimated)

PRIMARY OUTCOMES:
Change from baseline intraocular pressure at month 1 follow up | Baselines and month 1 follow up
  The intraocular pressure will be assessed by Goldmann Applanation Tonometry at baselines and month 1 follow up
Change from baseline intraocular pressure at month 3 follow up | Baselines and month 3 follow up
  The intraocular pressure will be assessed by Goldmann Applanation Tonometry at baselines and month 3 follow up
Change from baseline intraocular pressure at month 6 follow up | Baselines and month 6 follow up
  The intraocular pressure will be assessed by Goldmann Applanation Tonometry at baselines and month 6 follow up
Change from baseline intraocular pressure at month 12 follow up | Baselines and month 12 follow up
  The intraocular pressure will be assessed by Goldmann Applanation Tonometry at baselines and month 12 follow up

SECONDARY OUTCOMES:
The complete success rate at month 3 follow up | Month 3 follow up
  The complete success rate will be defined as intraocular pressure less than 18 mmHg with a 20 percent reduction without anti-glaucoma medication at month 3 follow up.
The complete success rate at month 1 follow up | Month 1 follow up
  The complete success rate will be defined as intraocular pressure less than 18 mmHg with a 20 percent reduction without anti-glaucoma medication at month 1 follow up.
The complete success rate at month 6 follow up | Month 6 follow up
  The complete success rate will be defined as intraocular pressure less than 18 mmHg with a 20 percent reduction without anti-glaucoma medication at month 6 follow up.
The complete success rate at month 12 follow up | Month 12 follow up
  The complete success rate will be defined as intraocular pressure less than 18 mmHg with a 20 percent reduction without anti-glaucoma medication at month 12 follow up.
The qualified success rate at month 3 follow up | Month 3 follow up
  The qualified success rate will be defined as intraocular pressure less than 18 mmHg with a 20 percent reduction with anti-glaucoma medication at month 3 followup.
The qualified success rate at month 6 follow up | Month 6 follow up
  The qualified success rate will be defined as intraocular pressure less than 18 mmHg with a 20 percent reduction with anti-glaucoma medication at month 6 followup.
The qualified success rate at the month 12 follow up | Month 12 follow up
  The qualified success rate will be defined as intraocular pressure less than 18 mmHg with a 20 percent reduction with anti-glaucoma medication at month 12 followup.
The qualified success rate at the month 1 follow up | Month 1 follow up
  The qualified success rate will be defined as intraocular pressure less than 18 mmHg with a 20 percent reduction with anti-glaucoma medication at month 1 followup.
Change from baseline the number of glaucoma medications at month 1 follow up | Baseline and month 1 follow up
  The number of glaucoma medications will be assessed at baseline and month 1 follow up.
Change from baseline the number of glaucoma medications at month 3 follow up | Baseline and month 3 follow up
  The number of glaucoma medications will be assessed at baseline and month 3 follow up.
Change from baseline the number of glaucoma medications at month 6 follow up | Baseline and month 6 follow up
  The number of glaucoma medications will be assessed at baseline and month 6 follow up.
Change from baseline the number of glaucoma medications at month 12 follow up | Baseline and month 12 follow up
  The number of glaucoma medications will be assessed at baseline and month 12 follow up.
Change from baseline the best-corrected visual acuity at month 6 follow up | Baseline and month 6 follow up
  The best-corrected visual acuity will be assessed using the Snellen chart at baseline and month 6 follow up.
Change from baseline the best-corrected visual acuity at month 12 follow up | Baseline and month 12 follow up
  The best-corrected visual acuity will be assessed using the Snellen chart at baseline and month 12 follow up.
Complications at month 1 follow up | Month 1 follow up
  The complications of surgery will be assessed at month 1 follow up.
Complications at month 3 follow up | Month 3 follow up
  The complications of surgery will be assessed at month 3 follow up.
Complications at month 6 follow up | Month 6 follow up
  The complications of surgery will be assessed at month 6 follow up.
Complications at month 12 follow up | Month 12 follow up
  The complications of surgery will be assessed at month 12 follow up.
Need to postoperative needling and laser goniopuncture at month 1 follow up | Month 1 follow up
  Need to postoperative needling and laser goniopuncture at month 1 follow up
Need to postoperative needling and laser goniopuncture at month 3 follow up | Month 3 follow up
  Need to postoperative needling and laser goniopuncture at month 3 follow up
Need to postoperative needling and laser goniopuncture at month 6 follow up | Month 6 follow up
  Need to postoperative needling and laser goniopuncture at month 6 follow up
Need to postoperative needling and laser goniopuncture at month 12 follow up | Month 12 follow up
  Need to postoperative needling and laser goniopuncture at month 12 follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No